CLINICAL TRIAL: NCT06449469
Title: Prospective Study on the Impact of Different Anti-thrombotic Therapies on Subclinical Leaflet Thickening and Its Temporal Dynamics in Transcatheter Bioprosthetic Aortic Valves (NOTION-4)
Brief Title: The Nordic Aortic Valve Intervention Trial 4 (NOTION-4)
Acronym: NOTION-4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Ole De Backer, Associate professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003361-19; 2020-003361-19 (EudraCT Number)
Record Dates: First submitted 2023-07-04; First posted 2024-06-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Valve Disease, Aortic
Keywords: heart valve disease; valvular bioprosthesis; aortic valve replacement; Randomized clinical trial; TAVI; Antitrombotic medication
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Diseases; Heart Valve Diseases; Aortic Valve Disease | interventions — Rivaroxaban; Aspirin; Clopidogrel; edoxaban; Dabigatran; apixaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinus rhythm - DOAC treatment (Experimental): Can either of the following anti-platelet components: dabigatran, apixaban, rivaroxaban, edoxaban or warfarin.
  Duration: 3 months, followed by an anti-platelet hereafter.
  Interventions: Drug: Rivaroxaban; Drug: Edoxaban; Drug: Dabigatran; Drug: Apixaban; Drug: Warfarin
- Sinus rhythm - Anti-platelet treatment (Active Comparator): Can be either of the following anti-platelet components: acetylsalicylic acid or clopidogrel.
  Duration: Lifelong
  Interventions: Drug: Acetylsalicylic acid; Drug: Clopidogrel

INTERVENTIONS:
Drug: Rivaroxaban — Direct oral anticoagulants (DOAC) treatment will encompass any of the approved drugs: Rivaroxaban, Edoxaban, Dabigatranetexilat, and Apixaban (Table 1). The DOAC dosage will be adjusted according to kidney function (Table 1) and may be adjusted during the study period according to potential changes in guideline recommendations or if new-onset AF would occur in the follow-up period. The specific DOAC prescribed will be determined by the treating physician. If the patient has already been prescribed Marevan before the aortic valve intervention, the patient will continue this medication following the procedure as an oral anticoagulant treatment, which is administered according to current guidelines.
  Other Names: SUB29263
  Arms: Sinus rhythm - DOAC treatment
Drug: Acetylsalicylic acid — Antiplatelets decrease platelet aggregation and inhibit thrombus formation. In NOTION-4 acetylsalicylic acid (75 mg once a day) is used as first line choice. For participants who are allergic to acetylsalicylic acid, clopidogrel (75 mg once a day) will be used. If the patient has already been prescribed Clopidogrel before the aortic valve intervention e.g. due to apoplexia, the patient will continue this medication following the procedure as an antiplatelet treatment, which is administered according to current guidelines.
  Other Names: SUB12730MIG
  Arms: Sinus rhythm - Anti-platelet treatment
Drug: Clopidogrel — Antiplatelets decrease platelet aggregation and inhibit thrombus formation. In NOTION-4 acetylsalicylic acid (75 mg once a day) is used as first line choice. For participants who are allergic to acetylsalicylic acid, clopidogrel (75 mg once a day) will be used. If the patient has already been prescribed Clopidogrel before the aortic valve intervention e.g. due to apoplexia, the patient will continue this medication following the procedure as an antiplatelet treatment, which is administered according to current guidelines.
  Other Names: SUB13395MIG
  Arms: Sinus rhythm - Anti-platelet treatment
Drug: Edoxaban — Direct oral anticoagulants (DOAC) treatment will encompass any of the approved drugs: Rivaroxaban, Edoxaban, Dabigatranetexilat, and Apixaban (Table 1). The DOAC dosage will be adjusted according to kidney function (Table 1) and may be adjusted during the study period according to potential changes in guideline recommendations or if new-onset AF would occur in the follow-up period. The specific DOAC prescribed will be determined by the treating physician. If the patient has already been prescribed Marevan before the aortic valve intervention, the patient will continue this medication following the procedure as an oral anticoagulant treatment, which is administered according to current guidelines.
  Other Names: SUB32701
  Arms: Sinus rhythm - DOAC treatment
Drug: Dabigatran — Direct oral anticoagulants (DOAC) treatment will encompass any of the approved drugs: Rivaroxaban, Edoxaban, Dabigatranetexilat, and Apixaban (Table 1). The DOAC dosage will be adjusted according to kidney function (Table 1) and may be adjusted during the study period according to potential changes in guideline recommendations or if new-onset AF would occur in the follow-up period. The specific DOAC prescribed will be determined by the treating physician. If the patient has already been prescribed Marevan before the aortic valve intervention, the patient will continue this medication following the procedure as an oral anticoagulant treatment, which is administered according to current guidelines.
  Other Names: SUB20521
  Arms: Sinus rhythm - DOAC treatment
Drug: Apixaban — Direct oral anticoagulants (DOAC) treatment will encompass any of the approved drugs: Rivaroxaban, Edoxaban, Dabigatranetexilat, and Apixaban (Table 1). The DOAC dosage will be adjusted according to kidney function (Table 1) and may be adjusted during the study period according to potential changes in guideline recommendations or if new-onset AF would occur in the follow-up period. The specific DOAC prescribed will be determined by the treating physician. If the patient has already been prescribed Marevan before the aortic valve intervention, the patient will continue this medication following the procedure as an oral anticoagulant treatment, which is administered according to current guidelines.
  Other Names: SUB25425
  Arms: Sinus rhythm - DOAC treatment
Drug: Warfarin — If the patient has already been prescribed Marevan before the aortic valve intervention, the patient will continue this medication following the procedure as an oral anticoagulant treatment, which is administered according to current guidelines.
  Other Names: SUB05128MIG
  Arms: Sinus rhythm - DOAC treatment

SUMMARY:
A randomized clinical trial investigating the incidence and temporal dynamics of subclinical leaflet thickening by cardiac CT in transcatheter bioprosthetic aortic valves in patients randomised to different anti-thrombotic strategies. Additionally, this study aims to examine a possible association between HALT and thromboembolic events.

DETAILED DESCRIPTION:
The NOTION-4 trial is an investigator-initiated, randomized, open label, comparative trial conducted at Rigshospitalet in Copenhagen and Skejby Sygehus in Aarhus. All adult patients that have undergone successful TAVI without contraindications for cardiac CT will be invited to participate in this study. Patients with SR and without known other indication for chronic OAC therapy will be randomized 1:1 either to lifelong ASA or to 3 months of DOAC followed by lifelong ASA. Patients with known AF will be randomized 1:1 to lifelong DOAC versus LAAC within 3 months followed by lifelong ASA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent successful TAVI according to Valve Academic Research Consortium (VARC)-2 criteria
* Residing in Denmark
* Provided written informed consent

Exclusion Criteria:

* Atrial fibrillation or any other indication for lifelong oral anticoagulant therapy
* Patient deemed not suitable for DOAC treatment because of previous life-threatening or major bleeding, e.g. intracranial haemorrhage or major gastrointestinal bleeding
* Patients with severe renal insufficiency (eGFR <30 mL/min/1.73 m2)
* Patient with absolute indication for anti-thrombotic therapy, e.g. recent PCI
* Iodine contrast allergy or other condition that prohibits CT imaging
* Age <18 years
* Women of childbearing potential, pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
HALT after 1 year | At 1 year after TAVI
  The number of patients with at least one prosthetic valve leaflet with HALT as assessed by cardiac CT at one year after TAVI.

SECONDARY OUTCOMES:
Combined clinical endpoint of all-cause mortality, thromboembolic event, and life-threatening or major bleeding | At 1 year and 5 years after TAVI
  Combined clinical endpoint of all-cause mortality, thromboembolic event, and life-threatening or major bleeding
Incidence of patients with HALT during follow up | At 3 months, 1 year and 5 years after TAVI
  The number of patients with at least one prosthetic valve leaflet with HALT as assessed by cardiac CT.
HALT on leaflets | At 3 months, 1 year and 5 years after TAVI
  Number of prosthetic leaflets with HALT at CT-scan.
Number of participants with ischemic stroke | At 3 months, 1 year and 5 years after TAVI
  The clinical endpoint of ischemic stroke verified by cerebrovascular imaging after the TAVI-procedure in patients with vs. without HALT.
Number of participants with stroke | At 3 months, 1 year and 5 years after TAVI
  Both ischemic and hemorrhagic strokes are included.
Number of participants with all-cause death | At 3 months, 1 year and 5 years after TAVI
  All cause mortality
Number of participants with cardiovascular mortality | At 3 months, 1 year and 5 years after TAVI
  Cardiovascular mortality as defined in current VARC definition
Number of participants with bleeding | At 3 months, 1 year and 5 years after TAVI
  Major bleeding or life-threatening bleeding
Number of participants with re-intervention | At 3 months, 1 year and 5 years after TAVI
  valve-in-valve TAVI, paravalvular leak closure, SAVR
Number of participants with aortic bioprosthetic dysfunction | At 3 months, 1 year and 5 years after TAVI
  According to EAPCI/ESC/EACTS definitions
Number of participants with bioprosthetic valve failure | At 3 months, 1 year and 5 years after TAVI
  Rate of failure according to EAPCI/ESC/EACTS definitions including Rate of valve-related deaths, re-intervention, severe hemodynamic SVD
NYHA classification | At 3 months, 1 year and 5 years after TAVI
  Assessing NYHA classification over time after TAVI
Quality of life scores with 5-level EQ-5D version (EQ5D-5L) | At 3 months, 1 year and 5 years after TAVI
  Assessing changes of quality of life scores after TAVI with 5-level EQ-5D version (EQ5D-5L) where lower scores mean better outcome (score from 1 to 5).
Quality of life scores with EQ Visual Analogue Scale (EQ VAS) | At 3 months, 1 year and 5 years after TAVI
  The EQ Visual Analogue Scale (EQ VAS) has minimum score 0 and maximum score 100, where higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ole De Backer, PhD, Principal Investigator — Rigshospital, Denmark
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Skejby, Aarhus
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thuraiaiyah J, Jorgensen TH, Jensen JM, Fuchs A, Willemen Y, Terkelsen CJ, Kofoed KF, Sondergaard L, Norgaard BL, De Backer O. Prospective study on the impact of different antithrombotic therapies on subclinical leaflet thickening and its temporal dynamics in transcatheter aortic valves-The NOTION-4 trial. Am Heart J. 2025 Jan;279:1-8. doi: 10.1016/j.ahj.2024.10.002. Epub 2024 Oct 5. PMID 39374638